CLINICAL TRIAL: NCT02653248
Title: Phase I Study of Stereotactic Body Radiation Therapy (SBRT) for Organ Confined Prostate Cancer
Brief Title: SBRT for Organ Confined Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Louis Potters, MD, Northwell Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-128B
Record Dates: First submitted 2015-08-26; First posted 2016-01-12 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Adenocarcinoma; Prostate Cancer
MeSH Terms: conditions — Adenocarcinoma; Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Patients will receive 5 fractions of Stereotactic Body Radiation Therapy (SBRT). Dose per fraction is 8Gy. Total Dose: 40Gy. To escalate the dose of stereotactic radiotherapy to a tumoricidal dose without exceeding the maximum tolerated dose in patients with organ confined prostate cancer.
  Interventions: Radiation: Stereotactic Body Radiation Therapy
- Cohort 2 (Experimental): Patients will receive 5 fractions of Stereotactic Body Radiation Therapy (SBRT). Dose per fraction is 9Gy. Total Dose: 45 Gy. To escalate the dose of stereotactic radiotherapy to a tumoricidal dose without exceeding the maximum tolerated dose in patients with organ confined prostate cancer.
  Interventions: Radiation: Stereotactic Body Radiation Therapy
- Cohort 3 (Experimental): Patients will receive 5 fractions of Stereotactic Body Radiation Therapy (SBRT). Dose per fraction is 10Gy. Total Dose: 50Gy. To escalate the dose of stereotactic radiotherapy to a tumoricidal dose without exceeding the maximum tolerated dose in patients with organ confined prostate cancer.
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — Patients will receive 5 fractions of SBRT radiation, treated every other day. No more than three fractions per week. Total dose will depend on cohort. Cohort 1: 40Gy, Cohort 2: 45 Gy, Cohort 3: 50 Gy.
  Other Names: SBRT

SUMMARY:
Stereotactic Body Radiation Therapy (SBRT) is a method of delivering radiation which can target the tumor more precisely and cause less damage to normal tissue. This is a Phase I research study looking at the safety of the dose of SBRT in organ confined prostate cancer.

DETAILED DESCRIPTION:
Radiation options for treating early stage prostate cancer can include external radiation therapy, which is radiation given outside the body, or prostate seed implant, which is placing radioactive seeds directly into the prostate. For external beam radiation therapy, treatment can last up to 9 weeks. Treatment is given daily, Monday through Friday. This may not be the most convenient option for some patients.

One way to potentially overcome this challenge is to deliver a more intense dose of radiation treatment to the tumor over a shorter amount of time. Stereotactic Body Radiation Therapy (SBRT) is a technique that treats the prostate with fewer treatments and can decrease the effect of radiation to the surrounding tissues. This study is a Phase I research study, which means that it will look at the safety of the dose of the SBRT. While SBRT itself is a standard of care method to administer radiation therapy, there has not been a specific dose outlined in the past. The aim of this study is to determine the dose that will treat the prostate cancer but cause the least amount of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable to provide informed consent
* Signed study specific informed consent
* Prostate specific-antigen (PSA) ≤ 10 Gleason 2-7
* Appropriate staging studies identifying as American Joint Committee on Cancer (AJCC) stage T1a, T1b, T1c, T2a, T2b
* No direct evidence of regional or distant metastases after appropriate staging studies
* Histologic confirmation of cancer by biopsy
* Age ≥ 18
* Karnofsky Performance Status must be ≥ 70
* American Urological Association (AUA) score must be ≤ 15 (alpha blockers allowed)

Exclusion Criteria:

* Female
* Positive lymph nodes of metastatic disease from prostate cancer
* Prior invasive malignancy unless disease free for a minimum of 3 years (carcinoma in situ of the breast, oral cavity, or non-melanomatous skin cancer are all permissable)
* T2c, T3, or T4 tumors
* Previous pelvic radiotherapy
* Previous surgery or chemotherapy for prostate cancer
* Previous transurethral resection of the prostate (TURP) or cryotherapy to the prostate
* Concomitant hormonal therapy
* Concomitant antineoplastic therapy (including surgery, cryotherapy, conventionally fractionated radiotherapy, and chemotherapy) while on this protocol
* History of Crohn's Disease or Ulcerative Colitis
* Previous significant obstructive symptoms; AUA score must be ≤ 15 (alpha blockers allowed)
* Significant psychiatric illness
* Severe, active co-morbidity defined as follows:
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months.
* Transmural myocardial infarction within the last 6 months
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
* Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol
* Acquired Immune Deficiency Syndrome (AIDS) based upon current Center Disease Control and Prevention (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
* History of treatment with potent immunosuppressive drugs for such conditions as post organ transplant, severe rheumatoid arthritis, etc. within the past 6 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-08; Primary Completion 2018-06 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 10 years
  Patients in each dose cohort will all be treated as a single dose group for dose escalation. Each cohort will have 7-15 patients. The study will be completed when either of the following events occur: 1- The Maximum Tolerated Dose (MTD) for a cohort is reached or 2- when the highest protocol dose level is treated and tolerated (10 Gy/fraction, total 50 Gy) where we consider the therapy likely to be tumoricidal per determination of the investigators. Follow up assessments will be: 1.5 months post treatment, 3, 6, 9, and 12 months post treatment, then every 6 months until five years post treatment, then annually for years 5-10. A period of 90 days must pass in order to assess toxicity. If 90 days have transpired without Dose Limiting Toxicity (DLT) in each of the first seven patients enrolled to a specific dose level, then dose escalation to the next level may proceed.

SECONDARY OUTCOMES:
Measurement of response - No Evidence of Disease | Up to 10 years
  No clinical evidence of disease on digital rectal examination.
Measurement of response - Equivocal Disease | Up to 10 years
  1. If abnormalities are present on the prostate digital rectal examination but are thought to be abnormal due to treatment and felt not to represent tumor.
  2. If clinical evidence of residual tumor is present but this has regressed from a previous examination.
Measurement of response - Radiographic Evidence of Disease | Up to 10 years
  1. Radiographic evidence of hematogenous (osseous, hepatic, etc.) and/or extrapelvic lymphatic of soft tissue relapse.
  2. Radiographic evidence of tumor recurrence within the pelvic lymphatics or soft tissue beneath the bifurcation of the common iliac arteries.
Time to Biochemical failure | Up to 10 years
  Prostate Specific Antigen (PSA) levels should be obtained per study calendar. The RTOG-ASTRO definition (also known as the Phoenix definition) of PSA failure will be used. Thus, when the PSA rises by more than 2 ng/ml above the lowest level (nadir) achieved after treatment, biochemical failure has occurred and the date of the failure is recorded at the time the nadir plus 2 ng/ml level is reached.
Disease-Free Interval | Up to 10 years
  The disease-free interval will be measured from the date of accession to the date of documentation of progression or until the date of death (from other causes).
Time to Distant Failure | Up to 10 years
  The time to distant failure will be measured from the date of study entry to the date of documented regional nodal recurrence or distant disease relapse. Patients with evidence of biochemical failure, but a negative prostate biopsy, will be considered as distant failure only.
Overall Survival | Up to 10 years
  The survival time will be measured from the date of accession to the date of death. All patients will be followed for survival. Every effort should be made to document the cause of death
Disease-Specific Survival | Up to 10 years
  Disease-specific survival will be measured from the date of study entry to the date of death due to prostate cancer. The following will be considered as failure events in assessing disease specific survival.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Potters, MD, Principal Investigator — North Shore-LIJ
Locations (1):
- North Shore-LIJ Cancer Institute, Lake Success, New York, United States

REFERENCES:
- [Derived] Potters L, Rana Z, Lee L, Cox BW. Outcomes of a Dose-Escalated Stereotactic Body Radiation Phase 1 Trial for Patients With Low- and Intermediate-Risk Prostate Cancer. Int J Radiat Oncol Biol Phys. 2019 Jun 1;104(2):334-342. doi: 10.1016/j.ijrobp.2019.01.092. Epub 2019 Feb 2. PMID 30721721